CLINICAL TRIAL: NCT06493669
Title: Study on the Correlation Between Treg Immune Cells on the Muscle Content and Cognitive Functions of the Elderly
Status: Recruiting | Type: Observational
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.LNBK.007
Record Dates: First submitted 2024-07-01; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Disorder Patients and Cognitive Assessment

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cognitive assessment — MoCA

SUMMARY:
In order to explore the impact of the level of the elderly Treg immune cells and the effects of different fat distribution and muscle content, the impact of the level of Treg immune cells on cognitive functions is explored. The correlation between visceral fat content, subcutaneous fat content and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

- aged 40-90 years old

Exclusion Criteria:

- previous diagnosis of dementia (including Alzheimer's disease, Lewy body dementia, Parkinson's disease, or other dementias) were excluded.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cognitive decline patient
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function decline | through study completion, an average of 1 year
  MoCA score <26

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT06493669/Prot_000.pdf